CLINICAL TRIAL: NCT01194999
Title: Evaluating the Change of Overactive Bladder Symptoms in Women Post Pubovaginal Sling Procedure for Stress Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barrie Urology Associates (Other)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Joseph Zadra, Chief of Urology, RVH, Barrie Urology Associates
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARC-2010-04
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Results first posted 2012-09-20 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-08

CONDITIONS: Urinary Bladder, Overactive
Keywords: OAB; Urinary Bladder, Overactive; Overactive Bladder Syndrome; VESIcare; Urgency; Nocturia; Frequency; Urge Urinary Incontinence; UUI; Pubovaginal Sling; PVS; Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Nocturia; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pubovaginal sling procedure (Experimental): Patients undergoing pubovaginal slings for stress urinary incontinence.
  Interventions: Device: Pubovaginal sling procedure

INTERVENTIONS:
Device: Pubovaginal sling procedure — The procedure involves placing a band of sling material directly under the bladder neck (ie, proximal urethra) or mid-urethra, which acts as a physical support to prevent bladder neck and urethral descent during physical activity. The sling also may augment the resting urethral closure pressure with increases in intra-abdominal pressure.

SUMMARY:
Pubovaginal sling (PVS) procedures are designed to curtail bladder leakage brought about by strenuous events such as child birth. A common purported side effect of PVS is urgency, the feeling of a compelling need to void with little warning. Other overactive bladder (OAB) adverse effects that some claim to develop post-op include further leakage (incontinence), frequency and nocturia (night time leakage). Anecdotal evidence from our clinic however, suggests that such de novo OAB symptoms are rarely induced by PVS, and may in fact be alleviated by said procedure. It is our aim to investigate this relationship in our clinic.

As a prospective member of this study, you will be asked to complete five surveys. The first survey will be administered prior to your pubovaginal sling. This will be used to establish your baseline experience of OAB. Over the course of the next year, you will be asked to complete the four remaining surveys at regularly scheduled check-ups.

ELIGIBILITY:
Inclusion Criteria.

* Post-pubovaginal sling patient.
* Complete agreement and signing of Informed Consent Form.

Exclusion Criteria.

* Currently taking antimuscarinics or α1 blockers.
* Patients with urinary retention, dependent on dialysis, gastroparesis or narrow angle glaucoma.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Zadra, MD CM FRCSC, Principal Investigator — Barrie Urology Associates - The Male/Female Health and Research Centre
Locations (1):
- Barrie Urology Associates - The Male/Female Health and Research Centre, Barrie, Ontario, Canada

REFERENCES:
- [Background] Toledo LG, Korkes F, Romero FR, Fernandes RC, Oliveira C, Perez MD. Bladder outlet obstruction after pubovaginal fascial sling. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Feb;20(2):201-5. doi: 10.1007/s00192-008-0759-8. Epub 2008 Nov 12. PMID 19002645
- [Background] Koch YK, Zimmern P. A critical overview of the evidence base for the contemporary surgical management of stress incontinence. Curr Opin Urol. 2008 Jul;18(4):370-6. doi: 10.1097/MOU.0b013e3282fdf8d5. PMID 18520757
- [Background] Chapple CR, Fianu-Jonsson A, Indig M, Khullar V, Rosa J, Scarpa RM, Mistry A, Wright DM, Bolodeoku J; STAR study group. Treatment outcomes in the STAR study: a subanalysis of solifenacin 5 mg and tolterodine ER 4 mg. Eur Urol. 2007 Oct;52(4):1195-203. doi: 10.1016/j.eururo.2007.05.027. Epub 2007 Jun 6. PMID 17574730
- [Background] Toglia MR, Ostergard DR, Appell RA, Andoh M, Fakhoury A, Hussain IF. Solifenacin for overactive bladder: secondary analysis of data from VENUS based on baseline continence status. Int Urogynecol J. 2010 Jul;21(7):847-54. doi: 10.1007/s00192-010-1120-6. Epub 2010 Mar 26. PMID 20339833
- [Background] Karram MM, Toglia MR, Serels SR, Andoh M, Fakhoury A, Forero-Schwanhaeuser S. Treatment with solifenacin increases warning time and improves symptoms of overactive bladder: results from VENUS, a randomized, double-blind, placebo-controlled trial. Urology. 2009 Jan;73(1):14-8. doi: 10.1016/j.urology.2008.08.485. Epub 2008 Nov 8. PMID 18995887

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred over the course of one year (October 2010 - October 2011). Patients requiring pubovaginal sling procedures for stress incontinence were invited to participate if they possessed limited comorbidities.
Pre-assignment Details: No significant pres-assignment measures were taken.
Period: Overall Study
Arm/Group | Pubovaginal Sling Procedure
Started | 132
Completed | 115
Not Completed | 17
Not completed — Lost to Follow-up | 17

BASELINE CHARACTERISTICS:
Arm/Group | Pubovaginal Sling Procedure
Number analyzed (Participants) | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 118
  >=65 years | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 51.35 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 132

OUTCOME MEASURES:

1. Primary Outcome: Change in OAB Symptoms Post Pubovaginal Sling Operation
Description: Measured through the administration of five overactive bladder questionnaires. Difference from baseline to follow-up evaluated using the Wilcoxon Signed Rank Test.
Time Frame: Baseline to final follow-up.
Population: All patients enrolled in the study were analyzed, except for those currently being treated with antimuscarinic therapy.
Measure: Number; unit: participants
Arm/Group | Pubovaginal Sling Procedure
Number analyzed (Participants) | 88
participants
  Patients with improved OAB | 63
  Patients with stable OAB | 21
  Patients with worsening OAB | 4
Statistical Analysis 1: Comparison: Pubovaginal Sling Procedure; Null hypothesis: No significant difference from baseline to final follow-up; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study.
Arm/Group | Pubovaginal Sling Procedure
Serious Adverse Events (participants affected / at risk) | 0/132
Other Adverse Events (participants affected / at risk) | 0/132

LIMITATIONS AND CAVEATS:
The V8 questionnaire used for patient surveying has been validated, but forms of such a nature present potential over and under reporting of symptoms. Loss to follow-up presents an issue, although we anticipate those lost experienced improvements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No